CLINICAL TRIAL: NCT02750085
Title: Evaluation of a Simple Pharmacokinetic Tool (myPKFiT™) to Guide Personalized Factor VIII Dosing in Patients With Hemophilia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Victor Blanchette (Other)
Collaborators: St. Paul's Hospital (Unknown); Montreal Children's Hospital of the MUHC (Other); Queen's University (Other); University Hospital, Motol (Other); The University Hospital Brno (Unknown); Royal Children's Hospital (Other); Sydney Children's Hospitals Network (Other); Royal Prince Alfred Hospital, Sydney, Australia (Other)
Responsible Party: Sponsor-Investigator, Victor Blanchette, Medical Director, Pediatric Thrombosis and Hemostasis Program, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Other Study IDs: myPKFiT™ Study
Record Dates: First submitted 2016-04-07; First posted 2016-04-25 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; pharmacokinetics; myPKFiT
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma collected from PK blood sampling
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 2-point and 6-point PK sampling

SUMMARY:
This is an investigator-initiated, industry-funded, multi-centre, international study that will be carried out prospectively at hemophilia treatment centres across Canada, the Czech Republic and Australia with SickKids as the coordinating site. The study will use a central laboratory not directly affiliated with any of the participating sites. Enrollment target is 50 participants, both adult and pediatric with severe hemophilia A receiving Advate, who will each complete a 2-point and 6-point pharmacokinetic (PK) sampling. The main aim is to compare the results of a 2 sample PK using clinically practical time points and myPKFiT™ (a web-based, population PK Bayesian tool) to a 6 sample population PK to determine whether the results obtained are in good agreement.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Hemophilia A;
* Severe disease (FVIII <2%);
* Receiving ADVATE for prevention of bleeding (prophylaxis) or receiving ADVATE on demand and a candidate for prophylaxis;
* Body weight ≤120 kg; and ≥12kg;

Exclusion Criteria:

* FVIII inhibitor positive (level of ≥0.6 Bethesda Units [BU] per mL using the Nijmegen modification of the Bethesda assay). Inhibitor status to be documented as negative prior to study enrollment according to the two most recent, consecutive inhibitor assays on record. If patients have < 50 exposure days, an assay will be completed centrally within a reasonable timeframe (approximately 8 weeks suggested) to make sure that they are negative.
* Body weight >120 kg or <12kg;
* Human immunodeficiency virus (HIV) positivity with cluster of differentiation 4 (CD4) count < 200 / microliter;
* Significant hepatic dysfunction, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 times upper limit of normal
* History of recent events that might affect FVIII half-life (e.g., infection, surgery or an invasive procedure) within 2 weeks of blood sampling.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe Hemophilia A
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Terminal half-life (t1/2) | 2 years
  2-point PK sampling protocol against 6-point PK sampling protocol
area under the plasma concentration versus time curve (AUC) | 2 years
  2-point PK sampling protocol against 6-point PK sampling protocol
Area under the moment curve (AUMC) | 2 years
  2-point PK sampling protocol against 6-point PK sampling protocol
In vivo recovery (IVR) | 2 years
  2-point PK sampling protocol against 6-point PK sampling protocol
Maximum concentration (Cmax) | 2 years
  2-point PK sampling protocol against 6-point PK sampling protocol
Clearance (Cl) | 2 years
  2-point PK sampling protocol against 6-point PK sampling protocol
Volume of distribution at steady state (Vss) | 2 years
  2-point PK sampling protocol against 6-point PK sampling protocol
Mean residence time (MRT) | 2 years
  2-point PK sampling protocol against 6-point PK sampling protocol
Time to factor VIII concentration of 1% over baseline | 2 years
  2-point PK sampling protocol against 6-point PK sampling protocol

CONTACTS AND LOCATIONS:
Overall Officials: Victor S Blanchette, MD, Principal Investigator — The Hospital for Sick Children

IPD SHARING:
Plan to Share IPD: No